CLINICAL TRIAL: NCT05770544
Title: DETERMINE (Determining Extended Therapeutic Indications for Existing Drugs in Rare Molecularly Defined Indications Using a National Evaluation Platform Trial): An Umbrella-Basket Platform Trial to Evaluate the Efficacy of Targeted Therapies in Rare Adult, Paediatric and Teenage/Young Adult (TYA) Cancers With Actionable Genomic Alterations, Including Common Cancers With Rare Actionable Alterations. Treatment Arm 03: Entrectinib in Adult, Paediatric and Teenage/Young Adult Patients With ROS1 Gene Fusion-Positive Cancers.
Brief Title: DETERMINE Trial Treatment Arm 03: Entrectinib in Adult, Paediatric and Teenage/Young Adult Patients With ROS1 Gene Fusion-Positive Cancers.
Acronym: DETERMINE
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Cancer Research UK (Other)
Collaborators: University of Manchester (Other); University of Birmingham (Other); Royal Marsden NHS Foundation Trust (Other); Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CRUKD/21/004 - Treatment Arm 3; IRAS ID: 1004057 (Other: IRAS)
Record Dates: First submitted 2023-02-22; First posted 2023-03-15 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Haematological Malignancy; Malignancy; Malignant Neoplasm; Lymphoproliferative Disorders; Neoplasms by Histologic Type; Neoplasms by Site; Cancer; Brain Neoplasms; Melanoma; Glioma; Solid Tumour
Keywords: Adult; Antineoplastic Agents; Cancer; Child; Entrectinib; Malignancy; Malignant Neoplasms; Molecular Targeted Therapy; Mutation; Neoplasms by Histologic Site; Neoplasms by Site; Oncogene; Paediatric; Protein Kinase Inhibitors; Rare; ROS1 Protein, human; Tumour-agnostic; Young adult
MeSH Terms: conditions — Hematologic Neoplasms; Neoplasms; Lymphoproliferative Disorders; Neoplasms by Histologic Type; Neoplasms by Site; Brain Neoplasms; Melanoma; Glioma | interventions — entrectinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment Arm 03 (Experimental): This entrectinib treatment arm is for adult, paediatric and TYA patients with ROS1 gene fusion-positive malignancies.
  Interventions: Drug: Entrectinib

INTERVENTIONS:
Drug: Entrectinib — Adult and paediatric patients with body surface area (BSA) ≥1.51 m^2 will receive entrectinib orally at a dose of 600 mg daily dose (three 200 mg capsules per day).
  Paediatric patients with BSA <1.51 m^2 will receive entrectinib at a dose of 100 mg (BSA=0.43-0.50 m^2) or 200 mg (BSA=0.51-0.80 m^2) or 300 mg (BSA=0.81-1.10 m^2) or 400 mg (BSA=1.11-1.50 m^2).
  Each cycle of treatment will consist of 28 days and patients may continue until disease progression without clinical benefit, unacceptable AEs or withdrawal of consent.
  Other Names: Rozlytrek

SUMMARY:
This clinical trial is looking at a drug called entrectinib. Entrectinib is approved as standard of care treatment for adult patients with non-small cell lung cancer (NSCLC) which have a particular molecular alteration called ROS1-positive, and patients 12 years old or above with solid tumours which have another type of change in the cancer cells. This means it has gone through clinical trials and been approved by the Medicines and Healthcare products Regulatory Agency (MHRA) in the UK.

Investigators now wish to find out if it will be useful in treating patients with other cancer types which have the same molecular alteration (ROS1-positive). If the results are positive, the study team will work with the NHS and the Cancer Drugs Fund to see if these drugs can be routinely accessed for patients in the future.

This trial is part of a trial programme called DETERMINE. The programme will also look at other anti-cancer drugs in the same way, through matching the drug to rare cancer types or ones with specific mutations.

DETAILED DESCRIPTION:
DETERMINE Treatment Arm 03 (entrectinib) aims to evaluate the efficacy of entrectinib in ROS1 gene fusion-positive rare* adult, paediatric and teenage/young adult (TYA) cancers and in common cancers where a ROS1 mutation or amplification is considered to be infrequent.

*Rare is defined generally as incidence less than 6 cases in 100,000 patients (includes paediatric and teenagers/young adult cancers) or common cancers with rare alterations.

This treatment arm has a target sample size of 30 evaluable patients. Sub-cohorts may be defined and further expanded to a target of 30 evaluable patients each.

The ultimate aim is to translate positive clinical findings to the NHS (Cancer Drugs Fund) to provide new treatment options for rare adult, paediatric and TYA cancers.

OUTLINE:

Pre-screening: The Molecular Tumour Board makes a treatment recommendation for the patient based on molecularly-defined cohorts.

Screening: Consenting patients undergo biopsy and collection of blood samples for research purposes.

Treatment: Patients will receive entrectinib until disease progression without clinical benefit, unacceptable adverse events (AEs) or withdrawal of consent. Patients will also undergo collection of blood samples at various intervals while receiving treatment and at the end of treatment visit (EoT).

After completion of study treatment, patients are followed up every 3 months for 2 years

THE DETERMINE TRIAL MASTER (SCREENING) PROTOCOL:

Please see DETERMINE Trial Master (Screening) Protocol record (NCT05722886) for information on the DETERMINE Trial Master Protocol and applicable documents.

ELIGIBILITY:
THE PATIENT MUST FULFIL THE ELIGIBILITY CRITERIA WITHIN THE DETERMINE MASTER PROTOCOL (NCT05722886) AND WITHIN THE TREATMENT ARM 03 (ENTRECTINIB) OUTLINED BELOW*

*When entrectinib-specific inclusion/exclusion criteria or precautions below differ from those specified in the Master Protocol, the entrectinib-specific criteria will take precedence.

Inclusion Criteria:

A. Confirmed diagnosis of a ROS1 gene fusion-positive malignancy, other than NSCLC, that has been identified using an analytically validated next-generation sequencing method.

B. Patients must be able and willing to undergo a fresh tissue biopsy at baseline and blood samples for translational research. Note that for patients with haematological malignancies or neuroblastomas, blood, bone marrow aspiration and/or trephine or lymph node biopsy samples may be taken.

C. Patients with a BSA of 0.43m^2 and over.

D. ADULT PATIENTS (≥18 years): Adequate organ function as per haematological and biochemical indices within the ranges defined in the protocol. These measurements should be performed to confirm the patient's eligibility.

E. PAEDIATRIC PATIENTS (<18 years): Adequate organ function as per haematological and biochemical indices within the ranges defined in the protocol. These measurements should be performed to confirm the patient's eligibility.

F. Women of childbearing potential are eligible provided that they meet the following criteria:

* Have a negative serum or urine pregnancy test before enrolment and either:
* Agree to use one form of highly effective birth control method such as:

I. Oral, intravaginal or transdermal combined (oestrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation

II. Oral, injectable or implantable progestogen-only hormonal contraception associated with inhibition of ovulation

III. Intrauterine device (IUD)

IV. Intrauterine hormone-releasing system (IUS)

V. Bilateral tubal occlusion

VI. Vasectomised partner

Plus a barrier method if using a hormonal method: male or female condom with or without spermicide; cap, diaphragm or sponge with spermicide OR

• Sexual abstinence;

Effective from the first administration of entrectinib, throughout the trial and for five weeks after the last administration of entrectinib.

G. Male patients with partners who are women of childbearing potential are eligible provided that they agree to the following, from the first administration of entrectinib, throughout the trial and for three months after the last administration of entrectinib:

* Agree to take measures not to father children by using a barrier method of contraception (condom plus spermicide) or to sexual abstinence.
* Non-vasectomised male patients with partners who are women of childbearing potential must also be willing to ensure that their partner uses a highly effective method of contraception as in F above.
* Male patients with pregnant or lactating partners must be advised to use barrier method contraception (e.g. condom) to prevent drug exposure of the foetus or neonate.

All male patients must refrain from donating sperm for the same period.

Exclusion Criteria:

A. Female patients who are pregnant, breastfeeding or planning to become pregnant during the trial or within five weeks following their last dose of entrectinib

B. Diagnosis of ROS1 fusion-positive NSCLC

C. Prior treatment with the same class of drug unless genetic profile demonstrates a mechanism of resistance known to be potentially sensitive to entrectinib

D. Patients with significant cardiovascular disease are excluded as defined by:

i. Current congestive heart failure requiring therapy (New York Heart Association III or IV) or known left ventricular ejection fraction (LVEF) <50% (moderate to severe).

ii. History of unstable angina pectoris or myocardial infarction up to three months prior to trial entry, or current poorly controlled angina (symptoms weekly or more).

iii. Presence of symptomatic or severe valvular heart disease (severe by local echo graphic criteria or American Heart Association/American Cardiac College Stage C or D).

iv. History of a clinically significant cardiac arrhythmia up to three months prior to trial entry (asymptomatic atrial fibrillation or asymptomatic first-degree heart block are permitted.

v. History of stroke (ischaemic or haemorrhagic) within the last three months.

• Patients with primary CNS tumours may be considered unless intra-tumoural bleeding has occurred within 2 weeks of the first dose of entrectinib, and patients with punctate CNS haemorrhages <3 mm may be considered.

E. Patients with a baseline QTcF (Corrected QT interval by Fridericia formula) interval longer than 450 milliseconds (ms) for male patients and 470 ms for female patients, patients with congenital long QTcF syndrome, and patients taking medicinal products that are known to prolong the QTc interval.

F. History of additional risk factors for Torsades de Pointes (e.g., family history of long QT syndrome)

G. Grade ≥2 peripheral neuropathy

H. Known active infections (bacterial, fungal or viral) that would interfere with the assessment of safety or efficacy of entrectinib, including human immunodeficiency virus (HIV) positivity. Patients with history of testing positive for HIV infection are eligible provided the each of the following conditions are met:

* CD4 count ≥350/μL;
* undetectable viral load;
* receiving antiretroviral therapy (ART) that does not interact with IMP (patients should be on established ART for at least four weeks); and
* no HIV/ acquired immune deficiency syndrome (AIDS)-associated opportunistic infection in the last 12 months.

I. Known hypersensitivity to entrectinib or any of the excipients

J. Patients who were administered a live, attenuated vaccine within 28 days prior to enrolment, or anticipation of need for such a vaccine during entrectinib treatment or within six months after the final dose of entrectinib

K. Patient unable to swallow entrectinib intact, without chewing, crushing or opening the capsules (as per the dosing schedule and suitable dosing strengths available). Any active gastrointestinal disease (e.g., Crohn's disease, ulcerative colitis, or short gut syndrome) or other malabsorption syndromes that would reasonably affect drug absorption

L. Patients with personal history of significant osteopenia (screening for osteopenia not required)

M. Any clinically significant concomitant disease or condition (or its treatment) that could interfere with the conduct of the trial or absorption of oral medications that would, in the opinion of the Investigator, pose an unacceptable risk to the patient in this trial

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-11-30 (Estimated); Primary Completion 2029-10 (Estimated); Study Completion 2029-10 (Estimated)

PRIMARY OUTCOMES:
Objective Response (OR) | Disease assessments to be performed up to 24 weeks from the start of trial treatment.
  An OR is defined as the confirmed occurrence of either a Complete Response (CR) or Partial Response (PR) according to Response Evaluation Criteria in Solid Tumours (RECIST) Version 1.1 criteria (or immune related [ir]-RECIST or standard imaging criteria for specific disease e.g. Response Evaluation in Neuro Oncology criteria [RANO]). In patients with leukaemia, OR will be defined as the occurrence of CR, CRi (CR with incomplete neutrophil recovery) or CRp (CR with incomplete platelet recovery). The trial will report the proportion of patients with an OR and 95% credible interval.
Durable Clinical Benefit (DCB) | Disease assessments to be performed up to 24 weeks from the start of trial treatment.
  DCB is defined as the absence of disease progression for at least 24 weeks from the start of trial treatment according to RECIST Version 1.1 criteria (or ir-RECIST or standard imaging criteria for specific disease e.g. RANO criteria) and, where relevant (e.g. for haematological malignancies), by standard bone marrow response assessment criteria. Alternative definitions of DCB based on different time points may be pre-specified for particular sub-cohorts if 24 weeks is not clinically relevant. The trial will report the proportion of patients with a DCB and 95% credible interval.

SECONDARY OUTCOMES:
Duration of response (DR) | Disease assessment every 2 cycles of entrectinib (each cycle is 28 days) and at EoT. After 24 weeks, it can be done every 12 weeks, on discussion with Sponsor. Follow-up visits are every 3 months after last dose of entrectinib for up to 2 years.
  DR is defined as the time from the date of the first confirmed CR or PR according to RECIST 1.1 (or ir-RECIST or standard imaging criteria for specific disease e.g. RANO criteria) to the date of disease progression. The trial will report the median DR and 95% credible interval.
Best percentage change in sum of target lesion / index lesion diameters (PCSD) | Disease assessment every 2 cycles of entrectinib (each cycle is 28 days) and at EoT. After 24 weeks, it can be done every 12 weeks, on discussion with Sponsor. Follow-up visits are every 3 months after last dose of entrectinib for up to 2 years.
  PCSD is defined as the greatest decrease or least increase in the sum of target lesion diameters (RECIST) or index lesion diameters (irRECIST) as a percentage compared to the baseline measurement. The trial will report the mean PCSD and 95% credible interval.
Time to treatment discontinuation (TTD) | From first dose of entrectinib to discontinuation of trial treatment up to 5 years.
  TTD is defined as the time from date of starting trial treatment to date of discontinuing trial treatment, in days estimated by the median of the posterior inverse gamma probability distribution. The trial will report the median TTD and 95% credible interval.
Progression-Free Survival time (PFS) | Disease assessment every 2 cycles of entrectinib (each cycle is 28 days) and at EoT. After 24 weeks, it can be done every 12 weeks, on discussion with Sponsor. Follow-up visits are every 3 months after last dose of entrectinib for up to 2 years.
  PFS is defined as the time from date of starting trial treatment to date of progression or date of death without a previous progression recorded estimated by the median of the posterior inverse gamma probability distribution.
Time to Progression (TTP) | Disease assessment every 2 cycles of entrectinib (each cycle is 28 days) and at EoT. After 24 weeks, it can be done every 12 weeks, on discussion with Sponsor. Follow-up visits are every 3 months after last dose of entrectinib for up to 2 years.
  TTP is defined as the time from date of starting trial treatment to date of progression or date of death without recorded progression censored rather than events. The trial will report the median TTP and 95% credible interval.
Growth Modulation Index (GMI) | Disease assessment every 2 cycles of entrectinib (each cycle is 28 days) and at EoT. After 24 weeks, it can be done every 12 weeks, on discussion with Sponsor. Follow-up visits are every 3 months after last dose of entrectinib for up to 2 years.
  GMI is defined as the ratio of TTP with the trial protocol treatment to TTP on the most recent prior line of therapy. The trial will report the mean GMI and 95% credible interval.
Overall Survival time (OS) | Time of death or up to 2 years after the EoT visit.
  OS is defined as the time from date of starting trial treatment to date of death from any cause estimated by the median of the posterior normal probability distribution.
Occurrence of at least one Suspected Unexpected Serious Adverse Reaction (SUSAR) | From the time of consent until 28 days after last dose of entrectinib (up to 5 years) or until patient starts another anti-cancer therapy, whichever came first. An average time frame will be presented with results entry.
  The trial will report the number of patients who experience at least one SUSAR to entrectinib.
Occurrence of at least one Grade 3, 4 or 5 entrectinib related AE | From the time of consent until 28 days after last dose of entrectinib (up to 5 years) or until patient starts another anti-cancer therapy, whichever came first. An average time frame will be presented with results entry.
  Number of patients who experience at least one entrectinib related Grade 3, 4 or 5 AE according to National Cancer Institute Common Terminology Criteria for Adverse Events Version 5.0.
EORTC-QLQ-C30 Standardised Area Under Summary Score Curve (QLQSAUC) in adult patients. | QoL surveys performed prior to inclusion, every cycle (each cycle is 28 days) and at EoT visit (up to 5 years).
  For adult populations, multiple measures of Quality of Life (QoL) will be generated from patient completion of the European Organisation for Research and Treatment of Cancer QLQ-C30 (EORTC-QLQ-C30) questionnaire (15 measures). For each patient the Summary Score from the questionnaire will be generated at each time point and the area under the curve generated by these scores over time will be calculated and standardised by the time frame. The trial will report the mean QLQSAUC and 95% credible interval.
EQ-5D Standardised Area Under Index Value Curve (EQ5DSAUC) in adult patients | QoL surveys performed prior to inclusion, every cycle (each cycle is 28 days) and at EoT visit (up to 5 years).
  For adult populations, two measures of QoL will be generated from patient completion of the EQ-5D-5L questionnaire. For each measure, scores based on responses from the questionnaire will be generated at each time point and the area under the curve generated by these scores over time will be calculated and standardised by the time frame. The trial will report the mean EQ5DSAUC and 95% credible interval.
Mean change from baseline in the PedsQL 4.0 Standardised Area Under total Scale Score Curve (PedsSAUC) in paediatric patients | QoL surveys performed prior to inclusion, every cycle (each cycle is 28 days) and at EoT visit (up to 5 years).
  For paediatric populations multiple measures of QoL will be generated from patient completion of the PedsQL 4.0 (4 measures and a Total Scale Score). The Summary Score from the questionnaire will be generated at each time point and the area under the curve generated by these scores over time will be calculated and standardised by the time frame. The trial will report the mean PedsSAUC and 95% credible interval.
Mean change from baseline in the PedsQL 4.0 Standardised Area Under total Scale Score Curve (PedsSAUC) in parents of paediatric patients | QoL surveys performed prior to inclusion, every cycle (each cycle is 28 days) and at EoT visit (up to 5 years).
  For paediatric populations multiple measures of QoL will be generated from patient's parent completion of the PedsQL 4.0 (4 measures). The Summary Score from the questionnaire will be generated at each time point and the area under the curve generated by these scores over time will be calculated and standardised by the time frame. The trial will report the mean PedsSAUC and 95% credible interval.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Krebs, Dr, Principal Investigator — The Christie Hospital
Locations (27):
- United Kingdom (27):
  - Belfast City Hospital, Belfast
  - University Hospital Birmingham, Birmingham
  - Birmingham Children's Hospital, Birmingham
  - Bristol Royal Hospital for Children, Bristol
  - Bristol Haematology and Oncology Centre, Bristol
  - Addenbrooke's Hospital, Cambridge
  - Velindre Cancer Centre, Cardiff
  - Cardiff Children's Hospital, Cardiff
  - Western General Hospital, Edinburgh
  - The Beatson Hospital, Glasgow
  - Royal Hospital for Children Glasgow, Glasgow
  - Leicester Royal Infirmary, Leicester
  - Alder Hey Hospital, Liverpool
  - University College London Hospital, London
  - Guy's Hospital, London
  - Great Ormond Street Hospital, London
  - Royal Manchester Children's Hospital, Manchester
  - The Christie Hospital, Manchester
  - Clatterbridge Cancer Centre, Metropolitan Borough of Wirral
  - Great North Children's Hospital, Newcastle
  - Freeman Hospital, Newcastle
  - Churchill Hospital, Oxford
  - John Radcliffe Hospital, Oxford
  - Weston Park Hospital, Sheffield
  - Sheffield's Children's Hospital, Sheffield
  - Southampton General Hospital, Southampton
  - The Royal Marsden Hospital, Sutton

IPD SHARING:
Plan to Share IPD: Yes
Individual de-identified patient data will be shared with researchers whose proposed use of the data is approved by a review committee of the Sponsor.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: All requests for data relating to this treatment arm that are made within 5 years from last patient last visit for the entrectinib treatment arm will be considered; requests made subsequently will be considered where possible.
Access Criteria: When a request has been approved, Cancer Research UK will provide access to the de-identified individual patient-level data and appropriate supporting information. A signed Data Sharing Agreement must be in place before accessing requested information. Requests should be submitted to drugdev@cancer.org.uk.

REFERENCES:
- See also: Overview of the DETERMINE trial — http://CRUK.org/determine
- See also: ClinicalTrials.gov record for DETERMINE Trial Master Screening Protocol (NCT05722886). — https://clinicaltrials.gov/ct2/show/NCT05722886